CLINICAL TRIAL: NCT05438849
Title: Improving Primary Care Understanding of Resources and Screening for Urinary Incontinence to Enhance Treatment
Brief Title: Improving Primary Care Access to Urinary Incontinence Treatment for Women Veterans
Acronym: PURSUIT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alayne D. Markland, Professor, University of Alabama at Birmingham
Other Study IDs: 1658917-2; U18HS028736 (AHRQ)
Record Dates: First submitted 2022-05-25; First posted 2022-06-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence
Keywords: women; Veterans; behavioral treatment; primary care
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women Veterans receiving primary care in VISN-7 of the VA Healthcare Administration (VHA): This project will include English-speaking, community-dwelling women Veterans 20 years or older with a diagnosis of UI (all types) and access to the internet via a mobile device or computer. Women Veterans who are currently pregnant or less than 12 weeks postpartum will be excluded. PURSUIT utilizes a mobile health application, called MyHealtheBladder, to connect patients with nonsurgical treatment options.
  Interventions: Behavioral: Mobile Health Application focused on behavioral treatments to treat urinary incontinence
- Health care providers in community-based outpatient clinics in VISN-7 of the the VHA: Community-Based Outpatient Clinics (CBOCs) from VA Integrated Service Network (VISN) 7 will be targeted, spanning the states of Alabama, Georgia, and South Carolina. VISN 7 CBOCs, serving at least 50 women Veterans with primary care services, will be recruited.
  Interventions: Combination Product: Practice Facilitation

INTERVENTIONS:
Behavioral: Mobile Health Application focused on behavioral treatments to treat urinary incontinence — Mobile health application for cell phones and computers that delivers evidence-based behavioral treatment for urinary incontinence, specifically tailored to women Veterans
  Other Names: MyHealtheBladder
  Groups: Women Veterans receiving primary care in VISN-7 of the VA Healthcare Administration (VHA)
Combination Product: Practice Facilitation — The toolkit has 4 components: (1) Practice Facilitation Visits, (2) Mobile-health or mHealth Application Training (MAT) training, (3) Access and education on the Data Dashboard, and (4) Health information technology (HIT) assistance.
  Other Names: Practice facilitation toolkit
  Groups: Health care providers in community-based outpatient clinics in VISN-7 of the the VHA

SUMMARY:
The PURSUIT project aims to improve access to evidence-based nonsurgical UI treatment for women Veterans in the Southeast region of the United States using the most effective remote delivery modality. Using cluster randomization, the study will compare two models at the practice level: (1) the use of a practice facilitation toolkit with a mHealth UI modality alone and (2) the practice facilitation toolkit with a mHealth UI model combined with education on clinical pathways for consultation. Patient level outcomes related to UI symptom improvement will be compared. Patient and provider perceptions of factors that could influence future remote UI treatment scalability will also be assessed. All primary care practices will receive practice facilitation with a PURSUIT toolkit that includes (1) 1-2 visits with a practice facilitator; (2) mobile-health or mHealth application training (MAT); 3) online resource hub; and (4) health information technology (HIT) assistance. PURSUIT's future goal is to disseminate the most effective modality for delivering nonsurgical UI treatment for women Veterans nationally within the VHA.

DETAILED DESCRIPTION:
PURSUIT aims to recruit 62 practices to participate in the trial implementation at 50 practices. Specifically, Community-Based Outpatient Clinics (CBOCs) from VA Integrated Service Network (VISN) 7 will be targeted, spanning the states of Alabama, Georgia, and South Carolina. The project will focus on VISN 7 CBOCs, serving at least 50 women Veterans with primary care services, will be recruited through connections with local women's health providers. The team estimates outreach to approximately 50,000 women Veterans and estimates that 30 percent (n=15,000) of these women will have UI symptoms, and, among those, 15 percent (n=2,500) will participate.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* English-speaking, community-dwelling women Veterans
* Diagnosis of UI (all types)
* Access to the internet via a mobile device or computer

Exclusion Criteria:

* Women Veterans who are currently pregnant or less than 12 weeks postpartum

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The team estimates outreach to approximately 50,000 women Veterans and estimates that 30 percent (n=15,000) of these women will have UI symptoms, and, among those, 15 percent (n=2,500) will participate.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence (UI) screening rates | Baseline and 6 months post-Baseline
  This will include measuring changes, over time, in UI diagnoses for women Veterans. These changes will be measured by pulling data on UI ICD-9 and ICD-10 codes collected via the program's clinical data dashboard.
Change, over time, in usage of the provider clinical data dashboard | Baseline and 6 months post-Baseline
  This will include capturing the unique number of clinic site "champions" (i.e. designated women's health provider) who engage with this program's clinical data dashboard. Dashboard engagement will be measured as the number of unique site champions who use the dashboard divided by the total number of site champions involved in this program.

SECONDARY OUTCOMES:
Enrollment rates of women Veterans for MyHealtheBladder | 2-, 4-, and 6-months post-Baseline
  Women receiving behavioral urinary incontinence treatment on MyHealtheBladder
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline and 2-months post-Baseline
  4-item tool to measure UI symptoms, scored on scale from 0-21 with a higher score indicating worse symptoms
Pelvic Floor Muscle Exercise (PFME) Adherence | 2-months post-Baseline
  2-item questionnaire to explore adherence to completing PFMEs
System Usability Scale | 2-months post-Baseline
  10-item questionnaire, using 5-point Likert scale, to gauge the usability of MHB. Scoring range is 0-100 with a higher score indicating the system is more usable,
Satisfaction and Perception of Improvement | 2-months post-Baseline
  3-item tool for feedback on participant satisfaction and perceived symptom improvement

CONTACTS AND LOCATIONS:
Overall Officials: Alayne D Markland, DO, MSc, Principal Investigator — UNIVERSITY OF ALABAMA AT BIRMINGHAM, BIRMINGHAM , AL
Locations (2):
- United States (2):
  - Birmingham VA Healthcare System, Birmingham, Alabama
  - Atlanta VA Health Care System, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goode PS, Markland AD, Echt KV, Slay L, Barnacastle S, Hale G, Wright MK, Lane TR, Burgio KL. A mobile telehealth program for behavioral treatment of urinary incontinence in women veterans: Development and pilot evaluation of MyHealtheBladder. Neurourol Urodyn. 2020 Jan;39(1):432-439. doi: 10.1002/nau.24226. Epub 2019 Nov 27. PMID 31774200

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT05438849/Prot_ICF_001.pdf